CLINICAL TRIAL: NCT04625998
Title: Systems Approach to Obesity Prevention in Underserved Children in Texas - Primary Prevention
Brief Title: Texas Childhood Obesity Research Demonstration (TX CORD) Project -Primary Prevention Study
Acronym: TXCORDPRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Baylor College of Medicine (Other); Seton Healthcare Family (Other); Texas Department of State Health Services (Other); Duke University (Other); City University of New York, School of Public Health (Other)
Responsible Party: Principal Investigator, Deanna Hoelscher, John P. McGovern Professor in Health Promotion & Director, Michael & Susan Dell Center for Healthy Living, UTSPH, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-11-0513 (Primary)
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Pediatric Obesity
Keywords: Pediatric obesity; Diet; Physical activity; Schools; Early care and education
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Elementary schools and Head Start centers in the intervention catchment areas implemented (1) an enhanced Coordinated Approach To Child Health (CATCH) program for elementary schools using the CATCH Coordination Guide (Enhanced CATCH Elementary School Program), and (2) CATCH Early Childhood program for Head Start Centers.
  Interventions: Behavioral: Enhanced CATCH Elementary School Program; Behavioral: CATCH Early Childhood (CEC)
- Comparison (No Intervention): Elementary schools and Head Start centers in the comparison catchment area used their regular school and early care and education (ECE) nutrition and physical activity programs. Elementary schools were required by law to implement a coordinated school health program.

INTERVENTIONS:
Behavioral: Enhanced CATCH Elementary School Program — Enhanced CATCH Elementary School Program is a Coordinated School Health Program that includes the CATCH Coordination Guide.
  Other Names: CATCH; Coordinated School Health Program
  Arms: Intervention
Behavioral: CATCH Early Childhood (CEC) — Implementation of the CATCH Early Childhood coordinated nutrition and physical activity program for Early Care and Education (ECE) centers.
  Other Names: CEC, CATCH EC
  Arms: Intervention

SUMMARY:
A systems approach emphasizes the linkage between individual behavior change strategies and social and physical environmental changes, which act synergistically to facilitate (or inhibit) healthy eating and active living. We hypothesize that among low income, ethnically diverse overweight and obese children, aged 2-12 years, a systems approach to child obesity will reduce BMI compared to primary prevention alone.

ELIGIBILITY:
Inclusion Criteria:

* Children attending selected elementary schools or Head Start Centers in the catchment areas.
* Ages 2 to 12

Exclusion Criteria:

* Children who are special needs

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4378 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Population-level Child Obesity as Defined by BMI z-score | 2 years
  Change in Body Mass Index z-score

CONTACTS AND LOCATIONS:
Overall Officials: Deanna M Hoelscher, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Nancy F Butte, PhD, Principal Investigator — Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoelscher DM, Butte NF, Barlow S, Vandewater EA, Sharma SV, Huang T, Finkelstein E, Pont S, Sacher P, Byrd-Williams C, Oluyomi AO, Durand C, Li L, Kelder SH. Incorporating primary and secondary prevention approaches to address childhood obesity prevention and treatment in a low-income, ethnically diverse population: study design and demographic data from the Texas Childhood Obesity Research Demonstration (TX CORD) study. Child Obes. 2015 Feb;11(1):71-91. doi: 10.1089/chi.2014.0084. Epub 2015 Jan 2. PMID 25555188
- [Background] Oluyomi AO, Byars A, Byrd-Williams C, Sharma SV, Durand C, Hoelscher DM, Butte NF, Kelder SH. The utility of Geographical Information Systems (GIS) in systems-oriented obesity intervention projects: the selection of comparable study sites for a quasi-experimental intervention design--TX CORD. Child Obes. 2015 Feb;11(1):58-70. doi: 10.1089/chi.2014.0054. Epub 2015 Jan 14. PMID 25587670